CLINICAL TRIAL: NCT06340854
Title: A Study to Evaluate the Efficacy and Safety of Once-weekly Insulin Icodec When Switching From Daily Basal Insulins Compared to Once-daily Insulin Glargine U100 in Adults With Type 2 Diabetes
Brief Title: A Research Study to See How Switching From a Daily Basal Insulin to a New Weekly Insulin, Insulin Icodec, Helps in Reducing the Blood Sugar Compared to Daily Insulin Glargine in Adults With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-7724; U1111-1292-6151 (Other: World Health Organization (WHO)); 2023-506084-34 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin icodec (Experimental): Participants will receive Insulin icodec subcutaneously once weekly.
  Interventions: Drug: Insulin icodec; Drug: Insulin glargine
- Insulin glargine U100 (Active Comparator): Participants will receive Insulin glargine subcutaneously once daily.
  Interventions: Drug: Insulin icodec; Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin icodec — Insulin Icodec will be administered subcutaneously.
Drug: Insulin glargine — Insulin glargine will be administered subcutaneously.

SUMMARY:
This study compares insulin icodec, a new insulin taken once a week, to insulin glargine, an insulin taken once a day. The study medicine will be investigated in participants with type 2 diabetes. Participants will either get insulin icodec or insulin glargine. Which treatment participants get is decided by chance. Insulin icodec is the new medicine being tested, while insulin glargine is already approved and can be prescribed by doctors. Participants will get one injection of insulin icodec once a week, or one injection of insulin glargine once a day, depending on the treatment group participants are assigned into. Participants will use a pen with a small needle to inject the medicine under participants skin into participants thigh, upper arm or stomach.The study will last for about 9 months, but participants will only be taking the study medicine for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D greater than equal to (≥) 180 days prior to the day of screening.
* HbA1c from 7.0-10.0% (53.0-85.8 mmol/mol), both inclusive, at screening confirmed by central laboratory analysis.
* Treated with once-daily or twice-daily basal insulin (Neutral Protamine Hagedorn insulin, insulin degludec, insulin detemir, insulin glargine 100 U/mL, or insulin glargine 300 U/mL) ≥ 90 days prior to the day of screening with or without any of the following anti-diabetic drugs/regimens with stable doses greater than equal to (≥) 90 days prior to screening: metformin, sulfonylureas, meglitinides (glinides), Dipeptidyl peptidase 4 (DPP-4) inhibitors, Sodium-Glucose Transport Protein 2 (SGLT2) inhibitors, thiazolidinediones, alphaglucosidase inhibitors, oral combination products (for the allowed individual oral anti- diabetic drugs), oral or injectable glucagon-like peptide 1 receptor agonists (GLP-1 RAs), injectable glucagon-like peptide 1(GLP-1)/ glucose-dependent insulinotropic polypeptide receptor agonist (GIP RA) combination products.
* Body mass index (BMI) ≤ 40.0 kilogram per square meter (kg/m^2).

Exclusion Criteria:

* Any episodes of diabetic ketoacidosis within 90 days prior to the day of screening.
* Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g., treatment with orlistat, thyroid hormones, or corticosteroids).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) | From baseline (week 0) to week 26
  Percentage point (%-point).

SECONDARY OUTCOMES:
Change in time in range 3.9-10.0 millimoles per litre (mmol/L) (70-180 milligrams per decilitre (mg/dL)) | From baseline (week -4 to 0) to week 22-26
  Percentage (%) of time.
Change in DTSQs (Diabetes Treatment Satisfaction Questionnaire status version) total treatment satisfaction | From baseline (week 0) to week 26
  DTSQs measures the satisfaction with diabetes treatment regimens in people with diabetes. The measure consists of 8 items, of which 6 items contributes to 1 global score. Higher scores on the global score indicate greater satisfaction with treatment. Global score ranges 0- 36. 6 items scored on a scale of 0 to 6. The higher the score the greater the satisfaction with treatment.
Number of severe hypoglycaemic episodes (level 3) | From baseline (week 0) to week 31
  Number of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (less than (<) 3.0 millimoles per litre (mmol/L) (54 mg/dL), confirmed by blood glucose (BG) meter) | From baseline (week 0) to week 31
  Number of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (<3.0 mmol/L (54 mg/dL),confirmed by BG meter) or severe hypoglycaemic episodes (level 3) | From baseline (week 0) to week 31
  Number of episodes.
Time spent < 3.0 mmol/L (54 mg/dL) | From week 22 to 26
  % of time.
Change in time spent > 10.0 mmol/L (180 mg/dL) | From baseline (week-4 to 0) to week 22-26
  % of time.
Mean weekly insulin dose | From week 24 to week 26
  Units (U).
Change in body weight | From baseline (week 0) to week 26
  Kilogram (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (70):
- United States (21):
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Clinical Trials Research, Lincoln, California
  - Northeast Research Institute of Florida, Fleming Island, Florida
  - South Broward Research LLC, Miramar, Florida
  - Endo Res Solutions Inc, Roswell, Georgia
  - Cotton-Oneill Diabetes and End, Topeka, Kansas
  - International Diabetes Center, Minneapolis, Minnesota
  - Jefferson City Medical Group, PC, Jefferson City, Missouri
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern NH Diabetes and Endo_Nashua, Nashua, New Hampshire
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare Wilmington, Wilmington, North Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Amarillo Medical Specialists, Amarillo, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Victorium Clinical Research, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Rainier Clin Res Ctr Inc, Renton, Washington
- Bulgaria (6):
  - "Medical Center Viva Feniks" Ood, Dobrich
  - MHAT "Knyaginya Klementina" -Sofia EAD, Sofia
  - UMHAT Aleksandrovska, Sofia
  - Medical Institute of Ministry of interior, Sofia
  - Medical centre Clinic Nova, Varna
  - Medical centre Berbatov Beli drin, Yambol
- Germany (6):
  - InnoDiab Forschung GmbH, Essen
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Institut für Diabetesforschung Osnabrück, Osnabrück
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- India (13):
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - Manipal Hospital, Old Airport Road, Bengaluru, Bengaluru, Karnataka
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry, Tamil Nadu
  - Gandhi Hospital & Medical college, Hyderabad, Telangana
  - Malla Reddy Narayana Multispeciality Hospital, Hyderabad, Telangana
  - Government Institute of Medical Sciences, Noida, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh, Chandigarh
  - Christian Medical College and Hospital, Ludhiana
- Japan (5):
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Tokyo Medical Univ. Hospital_Diabetes, Metabolism and Endocrinology, Shinjuku-ku, Tokyo, Tokyo
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Noritake Clinic, Ushiku-shi, Ibaraki
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole, Opole Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - NZOZ Vita-Diabetica Malgorzata Buraczyk, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Trialmed CRS, Piotrkow Trybunalski, Łódź Voivodeship
- Puerto Rico (2):
  - Advanced Clinical Research LLC, Bayamón
  - Manati Ctr For Clin Research, Manatí
- South Africa (6):
  - Hemant Makan, Johannesburg, Gauteng
  - Dr Moosa's Rooms, Lenasia, Gauteng
  - Botho ke Bontle Health Services, Pretoria, Gauteng
  - Dr A Amod, Durban, KwaZulu-Natal
  - Dr MB Moosa's Practice, Durban, KwaZulu-Natal
  - Dr Mahesh Duki Research And Trial Site, Durban, KwaZulu-Natal
- Spain (4):
  - Hospital Clinic i Provincial, Barcelona
  - ABS La Roca del Vallés, La Roca Del Vallés
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com